CLINICAL TRIAL: NCT04459663
Title: A Single-arm, Single-center, Phase II Clinical Study to Investigate the Efficacy and Safety of JS001 Combined With Axitinib in the Treatment of Advanced Non-small Cell Lung Cancer (NSCLC) With Negative Driving Gene After First-line Chemotherapy
Brief Title: JS001 Combination Therapy in NSCLC Negative Driving Gene After First-line Chemotherapy.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Li Zhang, MD (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, MD, Principal Investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS -149/JS001-ISS -CO49
Record Dates: First submitted 2020-06-27; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS001 combined with Axitinib (Experimental): JS001 combined with Axitinib in the treatment of advanced non-small cell lung cancer without activated EGFR mutation, ALK fusion and ROS fusion after or during first-line chemotherapy
  Interventions: Drug: Toripalimab injection combine with Axitinib

INTERVENTIONS:
Drug: Toripalimab injection combine with Axitinib — The patients in the group will be infused intravenously with fixed dose of 240mg JS001 on the first day of each cycle. Oral Axitinib 5mg bid (recommended interval of about 12 hours) was given daily from the second day of the initial cycle

SUMMARY:
This is a phase II, open, single-center clinical study to evaluate the efficacy and safety of JS001 combined with Axitinib in the treatment of advanced non-small cell lung cancer without activated EGFR mutation, ALK fusion and ROS fusion after or during first-line chemotherapy. About 50 subjects will be included in this study and will be treated with JS001 combined with acitinib. Each cycle is 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form (ICF);
2. Recurrent or advanced stage Ⅲ B or IV non-small cell lung cancer tested for EGFR mutation and ALK, ROS1 fusion gene, and all the driving gene was negative.
3. At least one measurable lesion (according to RECIST 1.1);
4. Failure of previous first-line standard chemotherapy:
5. Patients who agreed to provide previously stored tumor tissue specimens or fresh biopsies of tumor lesions
6. Age 18-75 years old, regardless of gender;
7. ECOG score 0-1;
8. Expected survival time ≥ 3 months;
9. Laboratory test value must show enough organ function

Exclusion Criteria:

1. Tumor histology or cytological pathology confirmed the presence of small cell lung cancer components, or sarcomatoid lesions;
2. Those who did not have a driving gene test;
3. Investigator believed that there was a clear bleeding tendency
4. Subjects who are currently participating in and receiving treatment in other studies, less than 4 weeks
5. Patients who had previously received second-line or more systemic chemotherapy for advanced NSCLC;
6. Patients who had received hematopoietic stimulating factors, within one week before the start of the study.
7. Uncontrollable or symptomatic hypercalcemia
8. Within 6 months before receiving the study treatment, they received chest (lung) radiotherapy > 30Gy, or received radiotherapy within 4 weeks or radiopharmaceuticals within 8 weeks, except for local palliative radiotherapy for bone metastases.
9. The adverse reactions of previous antineoplastic therapy have not yet recovered to CTCAE 5.0 grade ≤ 1 (except alopecia);
10. Major surgery or radiotherapy has been performed within 4 weeks before joining the group or has not yet fully recovered from the previous operation
11. Known active central nervous system (CNS) metastasis and / or cancerous meningitis;
12. Spinal cord compression without radical treatment of surgery and / or radiotherapy;
13. Uncontrolled tumor-related pain;
14. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage ;
15. Evidence of active pneumonia was found;
16. Clinically uncontrolled active infections;
17. Uncontrollable major seizures or superior vena cava syndrome;
18. Past or present co-existence of other malignant tumors;
19. Liver diseases known to be of clinical significance;
20. Those who have previously used any anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-CTLA-4 antibody and Axitinib;
21. Patients with active tuberculosis (TB);
22. Patients with any active autoimmune disease or history of autoimmune disease;
23. Any anti-infective vaccine;
24. Known (HIV) infection of human immunodeficiency virus;
25. The researchers believe that it can affect study compliance;
26. Patients who received systemic immunosuppressive drugs within the first 4 weeks of the first day of the first cycle;
27. History of severe allergy, anaphylaxis or other hypersensitivity to chimeric or humanized antibodies or fusion proteins;
28. Those who are known to be allergic to biological drugs;
29. Those who are known to be allergic to acitinib;
30. Patients with a history of arterial or venous thromboembolism;
31. Known hereditary or acquired bleeding and thrombotic tendencies;
32. Patients who have previously received allogeneic stem cell or parenchyma organ transplantation;
33. Pregnant or lactating women or women of childbearing age who were positive for serum pregnancy test before taking the drug for the first time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the antitumor activity of Toripalimab injection (JS001) combined with Axitinib | From date of randomization untiL intolerable toxicity, or investigators determined subjects could not benefit from the study treatment, or subjects withdrew their informed consent or died, or the the drug had been used continuously for 2 years.
  The objective tumor reponse rate ((ORR)) evaluated by the investigator based on the solid tumor efficacy evaluation criteria (RECIST 1.1)

SECONDARY OUTCOMES:
To evaluate the efficacy of JS001 combined with Axitinib | From date of randomization untiL intolerable toxicity, or investigators determined subjects could not benefit from the study treatment, or subjects withdrew their informed consent or died, or the the drug had been used continuously for 2 years.
  Duration of response, disease control rate, time to reponse, and progression free survival, overall survival, 6-month progression-free survival ,6-month and 1-year survival.
To evaluate the safety of JS001 combined with Axitinib | From date of randomization untiL intolerable toxicity, or investigators determined subjects could not benefit from the study treatment, or subjects withdrew their informed consent or died, or the the drug had been used continuously for 2 years.
  Overall incidence of adverse events (AE); The incidence of grade 3 or above AE; the incidence of severe adverse events (SAE); the incidence of drug-related AE; the incidence of AE resulting in permanent withdrawal of drugs; the incidence of AE leading to dose adjustment / suspension trial
To evaluate the correlation between programmed death receptor-ligand 1 (PD-L1) expression and anti-tumor response in tumor tissues. | From date of randomization untiL intolerable toxicity, or investigators determined subjects could not benefit from the study treatment, or subjects withdrew their informed consent or died, or the the drug had been used continuously for 2 years.
  To evaluate the changes of TBNK lymphocyte subsets and the correlation analysis of antitumor activity under the treatment of JS001 combined with acitinib tablets,and the possible predictive factors of curative effect by biomarker analysis, including but not limited to tumor tissue lymphocyte infiltration, PMBC, PD-L1, TMB (using NGS/WES method).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China